CLINICAL TRIAL: NCT06007144
Title: Unilateral Implantation of the SPIRION Laryngeal Pacemaker in Patients With Previous Permanent Glottal Enlargement
Brief Title: Performance of the SPIRION Laryngeal Pacemaker in BVFP Patients With Single-sided Glottal Enlargement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The DMC terminated trial GLP_2022C1P002 early, citing a no longer positive benefit risk ratio, very low recruitment (<1 patient/year/site), no added patient risk, but no relevant advantages to justify continuing the study and potential risks of TIVA.
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLP_2022CIP002; DRKS00032342 (Other: DRKS (Deutsches Register Klinischer Studien)); CIV-23-01-042030 (Other: EUDAMED)
Record Dates: First submitted 2023-07-26; First posted 2023-08-23 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Bilateral Vocal Cord Paralysis
Keywords: Bilateral Vocal Fold Paralysis; BVFP; Bilateral Vocal Cord Paralysis; BVCP; Laryngeal Pacemaker; Electrical Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): SPIRION Laryngeal Pacemaker System Implantation and follow-up
  Interventions: Device: SPIRION Laryngeal Pacemaker System Implantation and follow-up

INTERVENTIONS:
Device: SPIRION Laryngeal Pacemaker System Implantation and follow-up — Timeline of Visits
  * Screening
  * Baseline: Official baseline, assessment primary & secondary objectives
  * Implantation of device
  * Activation & fitting: Baseline active device; implanted device has just been activated; assessment of secondary objectives only
  * 8 FU Visits over 2 years after activation; Includes
    * Baseline Switch Off: results of the visit preceding a 14-day switch-off of the device; assessment of secondary objectives only
    * Endpoints for
      * Pivotal phase: 12 months after activation; official endpoint for assessment of primary & secondary objectives
      * Active post-pivotal phase: 24-month follow-up; endpoint for all secondary objectives
      * Switch Off: 2 Visits; assessment of secondary objectives only
    * Repeated checkpoints to assess device effects over 2 years: 5 visits; assessment of secondary objectives only
  Device shall increase respiratory patency during inspiration, assessed by normalized PIF; other outcome measures are used to assess secondary objectives

SUMMARY:
The goal of this clinical investigation is to learn about the use of a novel medical device, the SPIRION Laryngeal Pacemaker, in patients suffering from bilateral vocal fold paralysis (BVFP) and who have had at least one related surgery on one of their vocal folds. The main questions it aims to answer are:

* Is the use of the device safe?
* Does the device improve the participants ability to take a breath?

Participants will be implanted with the SPIRION Laryngeal Pacemaker and the development of their symptoms will be observed for the following 2 years.

DETAILED DESCRIPTION:
This clinical investigation aims to assess the long-term safety and performance of the SPIRION Laryngeal Pacemaker. The SPIRION Laryngeal Pacemaker is a new active implantable medical device designed and developed by MED-EL Elektromedizinische Geräte GmbH. It is currently in its pre-market approval phase and the results of this clinical investigation will be used to apply for EU market entry.

The SPIRION Laryngeal Pacemaker is intended to improve the symptoms of Bilateral Vocal Fold Paralysis (BVFP) patients with respiratory symptoms severe enough to require surgical treatment.

The SPIRION Laryngeal Pacemaker consists of 2 implantable (the SPIRION Electrode and the SPIRION Implant) and 1 external (the SPIRION Processor) components. The SPIRION Electrodes and the SPIRION Implant are placed subcutaneously in the neck and above the sternum, respectively. The SPIRION Processor is placed on the skin above the sternum.

The external SPIRION Processor transmits the stimulation parameters to the SPIRION Implant, which in turn transmits the stimulation via the SPIRION Electrode to the posterior cricoarytenoid muscle (PCA). The PCA stimulation induces the lateralization (abduction) of the respective vocal fold (VF) and thus increases the glottal gap and improves respiratory patency.

Each patient is foreseen to actively participate in this clinical investigation for a maximum of 28 months. Patients will be offered participation by their ear, nose, and throat specialist. In case a patient is interested, a thorough Informed consent process will be initiated. Patients will be tested for eligibility and if they pass, the baseline values regarding respiration, voice, and other symptoms will be recorded. A few days to weeks later, the SPIRION Laryngeal Pacemaker is implanted. The Implant is activated about 2 to 4 weeks after a successful implantation and is fitted to the individual needs of the patient. Subsequent follow-up (FU) visits are conducted after about 1, 3, 6, 9, 12, 18, and 24 months after the activation of the device. The results of the various tests meant to assesses the patients' quality of respiration, voice, and other symptoms are recorded. The SPIRION Laryngeal Pacemaker will be transiently deactivated twice between 12 and 24 months after activation. Tests will be performed in this period and compared with the previous and subsequent tests performed with the active device. In addition, patients' activity before implantation and during the 24-month FU period will be regularly assessed. Upon study conclusion, the patients will be actively followed-up every 6 months until the SPIRION Laryngeal Pacemaker receives a CE certification, or it is surgically removed.

The implantation of the SPIRION Laryngeal Pacemaker should generally improve the BVFP symptoms of patients regarding respiration, swallowing, and sleep quality. Voice quality should not be affected or even improve. Moderate physical activity (e.g., using an E-bike) should become possible, leading to an improved general quality of life.

Unlike surgical glottal enlargement, the implantation of the SPIRION Laryngeal Pacemaker should not lead to problems with swallowing and aspiration. In addition, it should lead to a lesser rate and /or severity of surgical complications and surgery-related side-effects.

ELIGIBILITY:
General information

The following patient categories can be recruited into this clinical investigation if they comply with all the selection criteria:

* Patients recruited in the previous first-in-human (FIH) clinical investigation 2011CIP001
* Patients with an open tracheostoma at the time of enrolment

Inclusion Criteria:

* Between 18 and 75 years old at the time of enrolment (i.e., informed consent form (ICF) signed)
* Diagnosed with BVFP for a minimum of 6 months
* Patients who underwent at least one permanent glottal enlargement. If revision surgeries were performed, they should have been conducted on the same side of the original surgery
* With sufficient autonomous respiratory capacity to maintain their vital functions independent of the SPIRION Laryngeal Pacemaker. Before a permanent closure of the tracheostomy is carried out during this clinical investigation, the Principal Investigator shall confirm that at least at rest, the failure of the SPIRION Laryngeal Pacemaker would not put the patient in a life-threatening condition because of insufficient respiratory patency
* The PCA innervating the vocal fold that never underwent a permanent glottal enlargement responds to electrical stimulation (clear abduction of the respective VF in response to electrical stimulation) within an Endoscopic Cap Electrode (ECE50) test
* Fluent in German.

Exclusion Criteria:

* Lack of compliance with any inclusion criteria
* Pregnant or breast-feeding women
* Patients suffering from an ongoing or chronic laryngeal inflammation at the time of enrolment
* Vocal fold immobility caused by arytenoid joint dysfunctions (e.g., arthritis, scarring, etc.), malignancies, central nervous system (CNS) pathologies, and/or systemic diseases
* Patients who underwent previous bilateral permanent surgical glottal enlargement
* Patients who never underwent a permanent glottal enlargement on either vocal fold
* Patients who underwent any other laryngeal surgeries (e.g., laryngeal framework surgery) that would compromise the correct SPIRION Electrode placement and/or the intended functionality of the SPIRION Laryngeal Pacemaker
* The adductor laryngeal muscles on either or both sides underwent a botulinum toxin injection that is still effective at the time of surgery (i.e., the respective VF position is either in intermediate or lateral position)
* Patients who underwent thoracic surgeries that would compromise at least one of the following procedures:

  * Correct placement of the SPIRION Electrode or SPIRION Implant
  * Connection of the SPIRION Implant with the SPIRION Electrode
  * Connection of the SPIRION Implant with the external SPIRION Processor
* Patients wearing an active implantable medical device at the time of enrolment
* Patients with a clinical history that would suggest a high probability that they would need an MRI
* Patients diagnosed with a malignant disease in the head and neck region
* Patients diagnosed with chronic airway infections or obstructions, or severe respiratory diseases (e.g., chronic obstructive pulmonary disease (COPD) grade II or higher)
* Patients who underwent external beam radiation therapy in the surgical area
* Patients diagnosed with a serious coagulation disorder requiring an uninterruptable use of anticoagulants
* Patients with known allergies to the SPIRION Laryngeal Pacemaker material in direct contact with the human body
* Patients suffering from moderate depression (Beck Depression Inventory II (BDI-II) ≥ 20) or any other psychological or psychiatric diseases
* Any anatomic, physiological, or medical conditions that may increase the risks linked to the SPIRION Laryngeal Pacemaker implantation and/or reduce its benefit for the patient
* Parallel participation in a device/drug clinical investigation in the period of data collection, which could confound the results of this clinical investigation
* Anything that, in the opinion of the Principal Investigator, would place the patient at increased risk or preclude the patient's full compliance with the general requirements of this clinical investigation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Device Safety | 12 Months
  Number of Adverse Events (AEs), Serious Adverse Device Effect (SADEs), and Device Deficiencies (DDs)
Device Performance - Respiration | 12 Months
  PIF (Peak Inspiratory Flow) [L/min]

SECONDARY OUTCOMES:
Voice Quality - Fundamental Frequency (F0) | 24 months
  F0 range [Hz]
Voice Quality - Sound Pressure Level (SPL) | 24 months
  SPL range [dB]
Voice Quality - Maximum Phonation Time (MPT) | 24 months
  MPT [s]
Voice Quality - Jitter | 24 months
  Jitter in percentage [%]
Voice Quality - Roughness, Breathiness, Hoarseness (RBH) | 24 months
  RBH - score between 0 and 3 for each characteristic, higher score indicates worse voice quality
Voice Quality - Dysphonia Severity Index (DSI) | 24 months
  DSI - calculated as 0,13 * MPT + 0,0053 * F0_maximal - 0,26 * SPL_minimal - 1,18 * Jitter + 12,4; the following ranges apply: abnormal voice (-5 < X ≤ 1,6); normal voice (1,6 < X ≤ 5), not evaluable (≤ -5)
Voice Quality - Voice Handicap Index (VHI)-9 | 24 months
  VHI-9 patient questionnaire - score between 0 and 36, higher score indicates worse voice quality)
Respiratory patency - Absolute Peak Expiratory Flow (PEF) | 24 months
  Absolute PEF [L/min]
Respiratory patency - Normalized PEF | 24 months
  Normalized PEF [L/min]
Respiratory patency - Absolute Peak Inspiratory Flow (PIF) | 24 months
  Absolute PIF [L/min]
Respiratory patency - Normalized PIF | 24 months
  Normalized PIF [L/min]
Respiratory patency - Absolute Vital Capacity (VC) | 24 months
  Absolute VC [L]
Respiratory patency - Normalized VC | 24 months
  Normalized VC [L]
Respiratory patency - Absolute Forced Expiratory Volume in one second (FEV1) | 24 months
  Absolute FEV1 [L]
Respiratory patency - Normalized FEV1 | 24 months
  Normalized FEV1 [L]
Respiratory patency - Absolute Forced Vital Capacity (FVC) | 24 months
  Absolute FVC [L]
Respiratory patency - Normalized FVC | 24 months
  Normalized FVC [L]
Respiratory patency - Tiffeneau Index | 24 months
  Tiffeneau Index - calculated as (FEV1/FVC)*100
Respiratory patency - Phonation quotient (PQ) | 24 months
  PQ - calculated as VC/MPT [L/s]
Respiratory patency - Estimated Mean Flow Rate (EMFR) | 24 months
  EMFR - calculated as 77+0.236*PQ
Respiratory patency - St. George's Respiratory Questionnaire (SGRQ) | 24 months
  SGRQ patient questionnaire - score between 0 and 100; higher score indicates worse health
Physical activity - 6 Minute Walk Test (6MWT) | 24 months
  6MWT [m]
Physical activity - Physical Activity Monitor (PAM) - Physical activity level (PAL) | 24 months
  PAL - calculated as Total Energy Expenditure [Kcal]/Basal Metabolic Rate[Kcal]
Physical activity - PAM - Activity/Rest durations | 24 months
  Durations of activity/inactivity/sleep measured in [h:m] and [%]
Physical activity - PAM - Movement intensity | 24 months
  Movement intensity [g]
Physical activity - PAM - Number of steps | 24 months
  Average Number of steps per 24 h
Physical activity - PAM - Times out of bed | 24 months
  Number of Times out of bed
Swallow quality | 24 months
  MD Anderson Dysphagia Inventory (MDADI) patient questionnaire - total score between 20 and 100, higher score indicates better day-to-day functioning
Sleep quality | 24 months
  Pittsburgh Sleep Quality Index (PSQI) patient questionnaire - score between 0 and 21; higher score indicates worse sleep quality
Participant's Quality of Life - Short Form-36 (SF-36) questionnaire | 24 months
  SF-36 patient questionnaire - score between 0 and 100, higher score indicates better health
Participant's Quality of Life - Glasgow Benefit Inventory (GBI) | 24 months
  GBI patient questionnaire - score between -100 and 100, negative scores indicate a poor outcome, positive scores indicate a good outcome
Symptoms | 24 months
  Symptom form - Log of symptoms and symptom severity during visits, descriptive evaluation
Symptoms and Patient Observations | 24 months
  Weekly Journal - Log of symptoms, symptom severity, and device use at home, descriptive evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Müller, Prof. Dr., Principal Investigator — SRH Wald-Klinikum Gera GmbH; Berit Schneider-Stickler, Prof. Dr., Principal Investigator — Medical University of Vienna; Dirk Mürbe, Prof. Dr., Principal Investigator — Charité - Medical University of Berlin; Claus Potoschnig, Univ-Doz.Dr., Principal Investigator — Tirol Kiniken GmbH; Jan-Constantin Kölmel, Dr., Principal Investigator — Stuttgart Hospital - Katharinenhospital; Rudolf Hagen, Prof. Dr.Dr., Principal Investigator — University Hospital of Würzburg
Locations (6):
- Austria (2):
  - Tirol Kliniken GmbH, Innsbruck, Tyrol
  - Medical University of Vienna, Vienna
- Germany (4):
  - Stuttgart Hospital - Katharinenhospital, Stuttgart, Baden-Wurttemberg
  - University Hospital of Würzburg, Würzburg, Bavaria
  - SRH Wald-Klinikum Gera GmbH, Gera, Thuringia
  - Charité - Medical University of Berlin, Berlin

IPD SHARING:
Plan to Share IPD: No